CLINICAL TRIAL: NCT05956483
Title: A Confirmatory Study of the Rapid Mood Screener for Bipolar 1 Disorder to Evaluate Capability to Distinguish Between Subjects With Unipolar Major Depressive Disorder and Bipolar 1 in a Real-world Setting
Brief Title: Study to Assess Accuracy of Rapid Mood Screener in Adult Participants With Unipolar Major Depressive Disorder or Bipolar 1 Disorder in Real World Setting
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H23-890
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder (BP1); Unipolar major depressive disorder (MDD); Rapid Mood Screener (RMS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rapid Mood Screener (RMS): Participants with Unipolar Major Depressive Disorder and Bipolar 1 Depression will be evaluated with RMS questionnaire and MINI interview.

SUMMARY:
Bipolar I Disorder (BP1)is a severe chronic mood disorder characterized by manic and depression. BP1 has high probability of being misunderstood as unipolar major depressive disorder (MDD). The purpose of this study is to confirm Rapid Mood Screener (RMS) effectively classifies participants with BP1.

Rapid Mood Screener (RMS) is a brief 6-item clinician-administered checklist, in which a participant's endorsement of four or more questions should trigger further clinical evaluation for BP1. Approximately 404 participants (303 with confirmed unipolar MDD and 101 with confirmed BP1) will be enrolled in the United States.

Participants will be answering RMS questionnaire and accuracy will be measured against Mini-International Neuropsychiatric Interview (MINI) interview.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to provider with primary complaint of new or continuing depressive symptoms.
* May be treatment naïve even if not in their first depressive episode.
* Meets one of the following criteria:

  * Previously treated and currently off medication.
  * Currently using an antidepressant, atypical antipsychotic for mood disorder, or mood stabilizer.

Exclusion Criteria:

* Hospitalized or admitted to the emergency room due to mental health issues in the past 30 days.
* Currently experiencing a manic episode.
* History of schizophrenia or depression due to another psychotic disorder or a medical, organic, or drug-induced cause or a neurocognitive disorder (dementia/delirium) (as defined by Diagnostic and Statistical Manual of Mental Disorders [DSM-V] criteria).
* Participant did not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Bipolar 1 Disorder or Unipolar Major Depressive Disorder
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) of Rapid Mood Screener (RMS) | Day 1
  PPV is defined as True Positive(TP)/(TP + False Positive (FP)).
Negative Predictive Value (NPV) of Rapid Mood Screener (RMS) | Day 1
  NPV is defined as True Negative(TN)/(TN + False Negative (FN)).
Sensitivity of Rapid Mood Screener (RMS) | Day 1
  Sensitivity is defined as TP/(TP+FN).
Specificity of Rapid Mood Screener (RMS) | Day 1
  Specificity is defined as TN/(TN+FP).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (9):
- United States (9):
  - ATP Clinical Research, Inc /ID# 255223, Costa Mesa, California
  - CT Clinical Research /ID# 253488, Cromwell, Connecticut
  - UHC Research /ID# 263151, Doral, Florida
  - J&A Clinical Research /ID# 263034, Doral, Florida
  - MedOne Clinical Research /ID# 263031, Miami, Florida
  - Oceanic Research Group /ID# 263032, North Miami Beach, Florida
  - Health Synergy Clinical Research LLC /ID# 262998, Okeechobee, Florida
  - Interventional Psychiatry of Tampa Bay /ID# 253526, Tampa, Florida
  - Richard Louis Price, M.D., LLC /ID# 253527, Monsey, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H23-890